CLINICAL TRIAL: NCT04675671
Title: Analgesic and Anxiety Efficacy of Preemptive Pregabalin Administration in Arthroscopic Shoulder Surgery: a Prospective Randomized Controlled Trial
Brief Title: Analgesic and Anxiety Efficacy of Preemptive Pregabalin
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, Principal investigator, Selcuk University
Other Study IDs: farukcicekci4
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Analgesia; Anxiety; Arthroscopic Shoulder Surgery
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregabalin group (Group P): Group pregabalin patients will be received 75 mg of pregabalin twice daily for 2 days before surgery
  Interventions: Other: Preoperative and postoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-S)] and [ Spielberg's State-Trait Anxiety Inventory (STAI-T) ]
- Control group (Group C): The Control group will be received plasebo capsule mg at the same point in time
  Interventions: Other: Preoperative and postoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-S)] and [ Spielberg's State-Trait Anxiety Inventory (STAI-T) ]

INTERVENTIONS:
Other: Preoperative and postoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-S)] and [ Spielberg's State-Trait Anxiety Inventory (STAI-T) ] — The postoperative pain is measured and evaluated by Visual Analog Scale (VAS= 0 = no pain to 10 = worst pain)
  Other Names: postoperative pain

SUMMARY:
Effective postoperative pain control after arthroscopic shoulder surgery optimizes postoperative rehabilitation, reduces anxiety, and can increase patient satisfaction and postoperative healing by providing amnesia and sedation. Few literature is available for postoperative pain management, including intra-articular local anesthetic infiltration, regional nerve blocks, patient-controlled analgesia (PCA) with intravenous opioid, and oral nonsteroidal anti-inflammatory and gabapentinoid drugs. Recently, gabapentinoides such as pregabalin have also shown to have potential in the treatment of acute postoperative pain as part of multimodal analgesia, due to their possible opioid consumption-reducing effects and prevention of post-surgical chronic pain. Pregabalin is an anticonvulsant drug that reduces calcium entry into the nerve terminals of the central nerve and also reduces levels of substance P, glutamate and noradrenaline, all of which play a major role in creating a feeling of pain. It is well known that pregabalin reduces central sensitization and hyperalgesia after tissue injury by inhibiting calcium influx in voltage-gated calcium channels. These theoretical advantages have led to clinical trials to confirm the analgesic effectiveness of oral pregabalin for postoperative pain management in various surgical procedures.

DETAILED DESCRIPTION:
One day before the scheduled surgery, a staff who was not included in this study will assign patients to the random Pregabalin group (n = 30) and the Control group (n = 30) according to a will be computerized randomization table. The hospital pharmacy will prepare all medications in same capsules, and all the medications of study drug will performe by a nurse, who was not involved in other process of this study administered the capsules orally with sips of water. Group pregabalin patients will receive 75 mg of pregabalin twice daily for 2 days before surgery. the Control group will receive plasebo capsule mg at the same point in time. The last doses one hour before induction of anesthesia. The double-blind design in this study included blinding of anesthesiologist, orthopedic surgeon, nurse giving the drugs, and the patients.

No other sedative premedication will be given to all patients. Anesthesia will induce with propofol 2 mg.kg-1and remifentanil 0.5-1 µg.kg-1, and tracheal intubation will facilitate with rocuronium 0.6 mg.kg-1. Anesthesia will maintaine with a continuous infusion of remifentanil 0.05-0.2 µg.kg-1.min-1 and sevoflurane 2-2.5 vol% to maintain a bispectral index scale (BIS) values of 40 to 60. All surgeries will be performed by an experienced orthopedic surgeon. At the end of the surgery, sevoflurane and remifentanil will stop and residual neuromuscular paralysis will antagonize, and extubation will performe when the patient had sufficient expiration. Age, gender, body mass index, the duration of anesthesia surgery and the type of surgery will record. In the preoperative period, and duration of operation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiologists (ASA) grade I or II
* Aged 18-65 years
* Scheduled for elective Arthroscopic shoulder surgery (Bankart or rotator cuff repair)

Exclusion Criteria:

* Major neurological, cardiovascular, metabolic, respiratory, renal disease or coagulation abnormalities
* Body mass index over 40 kg / m2
* Chronic alcohol and substance use
* History of upper gastrointestinal bleeding or perforation
* Using more than 5 mg / day of oral morphine or equivalent opioids (more than 1 month)
* Patients who are allergic to the drugs used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be scheduled patients of American society of Anesthesiologists (ASA) grade I or II, aged 18-65 years, and scheduled for elective Arthroscopic shoulder surgery (Bankart or rotator cuff repair) under general anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-03-03 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-S)] | Preoperatif 4 hours before
  STAI-S consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Preoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-T)] | Preoperatif 4 hours before
  STAI-T consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Preoperative anxiety measurement [Spielberger's State Anxiety Scale (STAI-S) | postoperative within 24 hours
  STAI-S consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
The postoperative pain will be measured by Visual Analog Scale (VAS) | postoperative within 24 hours
  Visual Analog Scale will be evaluated between VAS= 0 (no pain) and VAS=10 levels (worst pain).This parameter is measured from 10mins, 30 mins, 1 hour, 3 hours, 6 hours, 12 hours and 24 hours post-operatively,

SECONDARY OUTCOMES:
The time to first requirement for analgesia is the second outcome. | 48 hours
  It will be measured within 48 hours postoperatively
The total amount of morphine consumed | 48 hours
  It will be measured within 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, School of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided